CLINICAL TRIAL: NCT05592262
Title: A Randomized, Open-label, Single-dose, Two-cycle, Two-sequence, Cross-controlled Study Evaluating the Pharmacokinetic Effects of a High-fat Diet on Oral Administration of SHR2554 Tablets in Healthy Adult Subjects in China
Brief Title: Pharmacokinetic Test of High-fat Diet After Oral Administration of SHR2554 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR2554-I-109
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, single-dose, two-cycle, two-sequence, cross-controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR2554
- Treatment group B (Experimental)
  Interventions: Drug: SHR2554

INTERVENTIONS:
Drug: SHR2554 — On an empty stomach - after meals
  Arms: Treatment group A
Drug: SHR2554 — After meals - on an empty stomach
  Arms: Treatment group B

SUMMARY:
The objective of the study is to assess the effect of food on the pharmacokinetics, and safety of SHR2554 Tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged between 18 and 45 (inclusive) at the time of signing the informed consent;
2. Body weight ≥ 50.0 kg for men and body weight ≥ 45.0 kg for women, and body mass index (BMI) within the range of 19.0 to 26.0 kg /m2 (inclusive);
3. The mean value of three 12-lead ECG tests was normal or abnormal but not clinically significant, the time limit from Q wave to T wave was < 430 msec for male (QTcF), and < 450 msec for female (QTcF), and the heart rate was in the normal range or abnormal but not clinically significant.
4. Creatinine clearance (CLCr) ≥80 mL/min, and creatinine is less than or equal to the upper limit of normal value;
5. Participants should have no fertility plan from signing the informed consent until 6 months after the last medication, take effective contraceptive measures voluntarily and have no sperm donation plan. The serum HCG test of fertile women must be negative before Screening;
6. Participants should sign the informed consent before the study, and fully understand the content, process and possible adverse reactions of the study.

Exclusion Criteria:

1. Patients with abnormal vital signs (systolic blood pressure <90 mmHg or >140 mmHg, diastolic blood pressure <50 mmHg or >90 mmHg) or abnormal physical examination, laboratory examination (blood routine, blood biochemistry, urine routine, coagulation function), 12-lead electrocardiogram and other tests with clinical significance;
2. Abnormal X-ray examination with clinical significance;
3. Hepatitis B surface antigen, hepatitis C antibody and treponema pallidum antibody are positive or HIV antibody is not negative;
4. Allergic constitution, including history of severe drug allergy or drug allergy; Allergic history to SHR2554 tablets or the excipients thereof;
5. Previous history of cardiovascular diseases such as myocarditis, coronary heart disease, pathological arrhythmia, stroke, etc.;
6. Lung diseases, including invasive lung disease, pneumonia, dyspnea, etc.;
7. History of chronic kidney disease, renal insufficiency, and renal anemia;
8. History of dysphagia or any gastrointestinal disease that affects drug absorption;
9. Any uncontrolled peptic ulcer, colitis, pancreatitis, etc.;
10. Other important organs of primary diseases, such as the nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism, and clear history of musculoskeletal system including but not limited to tumor patient or a history of cancer, such as not good control of diabetes, high blood pressure, etc.), the researchers think that don't fit for the researchers;
11. Patients who had undergone any surgery that would affect drug absorption, distribution, metabolism, or excretion within 3 months prior to screening;
12. Took hepatotoxic drugs (e.g. Dapsone, erythromycin, fluconazole, ketoconazole, rifampin) within 6 months before screening;
13. Candidates who participated in clinical trials within 3 months before screening;
14. Took any drug that alters the activity of liver enzymes within 28 days prior to taking the study drug;
15. Took any prescription or over-the-counter medications in the 7 days prior to taking the study drug;
16. Took any vitamin products or herbs in the 7 days prior to taking the study drug;
17. History of substance abuse, drug use and/or alcohol abuse: a history of substance abuse in the 6 months prior to screening, or a positive urine substance abuse screening test in the screening/baseline period, or drug use in the 3 months prior to screening; Heavy drinkers (14 units of alcohol per week: 1 unit = 285mL beer, 25mL liquor, or 100mL wine; Smoking ≥5 cigarettes per day), or having a positive alcohol breath test during the screening period/baseline, or being unable to smoke or abstain during the trial;
18. Drinking grapefruit juice, beverages containing xanthine, caffeine, alcohol, strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, excretion within 48 hours before taking the study drug;
19. Participants who donated blood ≥400 mL or lost blood ≥400 mL within 3 months before screening, or received blood transfusion;
20. Patients with a history of needle sickness and blood sickness have difficulty in blood collection or cannot tolerate venipuncture blood collection;
21. Other factors considered by the investigator to be inappropriate for trial participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of SHR2554: Cmax | day 1 to day 10
Pharmacokinetic parameters of SHR2554: AUC0-t | day 1 to day 10
Pharmacokinetic parameters of SHR2554: AUC0-∞ (if applicable) | day 1 to day 10

SECONDARY OUTCOMES:
Pharmacokinetic parameters of SHR2554: Tmax | day 1 to day 10
Pharmacokinetic parameters of SHR2554: t1/2 | day 1 to day 10
Pharmacokinetic parameters of SHR2554: CL/F | day 1 to day 10
Pharmacokinetic parameters of SHR2554: Vz/F | day 1 to day 10
The incidence and severity of adverse events/serious adverse events. | from ICF signing date to approximate day 17

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided